CLINICAL TRIAL: NCT00910858
Title: A Pharmacokinetic And Pharmacodynamic Study Of Oral Lenalidomide (Revlimid) In Subjects With Low- Or Intermediate-1-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-PK-002; NCT00360880 (obsolete NCT alias)
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Low- or Intermediate-1-risk Myelodysplastic Syndrome (MDS)
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mg Lenalidomide (Experimental): Participants in the Pharmacokinetic Phase received a single 10 mg oral dose of lenalidomide on Day -7. During the Monotherapy Phase participants received 10 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  During the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg lenalidomide in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
  Interventions: Drug: Lenalidomide; Drug: Recombinant human erythropoietin
- 15 mg Lenalidomide Non-del 5q (Experimental): Following the enrollment of the first 25 patients into the Monotherapy Phase, a second group of 15 patients with low- or intermediate-1-risk MDS not associated with a del 5q (non-del 5q) cytogenetic abnormality were enrolled to receive 15 mg of lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure. During the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 15 mg lenalidomide in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
  Interventions: Drug: Lenalidomide; Drug: Recombinant human erythropoietin

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 5-mg capsules for oral administration
  Other Names: Revlimid
Drug: Recombinant human erythropoietin — Recombinant human erythropoietin (rhu-EPO) subcutaneous injection of 40,000 units.

SUMMARY:
The purpose of this study is to assess pharmacokinetic and pharmacodynamic characteristics of oral lenalidomide monotherapy administered to patients with Low- or Intermediate-1-risk Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Age ≥18 years at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Documented diagnosis of MDS that meets International Prognostic Scoring System (IPSS) criteria for Low- to Intermediate-1-risk disease.

   •Must have a diagnosis of low- or intermediate- risk MDS without a del 5q chromosomal abnormality (patients taking 15 mg starting dose only).
5. Must be able to provide adequate bone marrow (BM) aspirate and biopsy specimens for histopathological analysis and standard cytogenetic analysis during the screening procedure.
6. Red blood cell (RBC) transfusion-dependent anemia defined as having received ≥4 transfusions of RBCs within 56 days of randomization or symptomatic anemia (hemoglobin < 9.0 g/dl).
7. Failed prior treatment with recombinant human erythropoietin (rhu-EPO) (≥ 30,000 U/week x 6) or serum erythropoietin (EPO) concentration ≥500 mU/ml (hemoglobin < 9.0 g/dl).
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
9. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device [IUD], hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods, if needed.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Prior therapy with lenalidomide.
3. Proliferative white blood cell (WBC) ≥12,000/µL) chronic myelomonocytic leukemia (CMML).
4. MDS secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases.
5. Any of the following lab abnormalities:

   * Absolute neutrophil count (ANC) <500 cells/µL (0.5 x 10^9/L)
   * Platelet count <50,000/µL (50 x 10^9/L)
   * Serum creatinine > upper limit of normal (ULN)
   * Serum glutamic oxaloacetic transaminase/aspartate transaminase (SGOT/AST) or serum glutamic pyruvic transaminase/alanine transaminase (SGPT/ALT) >2.0 x ULN
   * Serum total bilirubin >2.0 mg/dL (34 µmol/L)
6. Prior ≥grade-2 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) allergic reaction to thalidomide.
7. Prior desquamating (blistering) rash while taking thalidomide.
8. Patients with ≥grade-2 neuropathy.
9. Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding.
10. Use of cytotoxic chemotherapeutic agents, erythropoietin, or experimental agents (agents that are not commercially available) for the treatment of MDS within 28 days of the first day of study drug treatment.
11. Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥3 years.
12. Any serious medical condition or psychiatric illness that will prevent the patient from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study.
13. Known human immunodeficiency virus (HIV-1) positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Komrokji RS, Lancet JE, Swern AS, Chen N, Paleveda J, Lush R, Saba HI, List AF. Combined treatment with lenalidomide and epoetin alfa in lower-risk patients with myelodysplastic syndrome. Blood. 2012 Oct 25;120(17):3419-24. doi: 10.1182/blood-2012-03-415661. Epub 2012 Aug 30. PMID 22936658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants were enrolled at 1 site in this study, with 12 participants enrolled in the Pharmacokinetic (PK) Phase of the study, 39 participants enrolled in the Monotherapy Phase of the study, and 23 participants enrolled in the Combined Treatment Phase of the study.
Pre-assignment Details: The Monotherapy Phase included an initial group of 24 patients (11 from the PK Phase and 13 newly enrolled) who participated in the multiple-dose PK assessment and a second group of 15 patients (15 mg Non-del 5q) for whom no PK samples were taken. Erythroid nonresponders or responders who relapsed could participate in the Combined Treatment Phase.
Groups:
- 10 mg Non-del 5q: Participants with low- or intermediate-1-risk myelodysplastic syndromes (MDS) not associated with a deletion 5q (del 5q) cytogenetic abnormality received a single 10 mg oral dose of lenalidomide on Day -7 in the Pharmacokinetic Phase.
  During the Monotherapy Phase participants received 10 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
- 15 mg Non-del 5q: Participants with low- or intermediate-1-risk MDS not associated with a deletion 5q (del 5q) cytogenetic abnormality were enrolled directly into the Monotherapy Phase and received 15 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 15 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
- 10 mg Del 5q: Participants with a deletion 5q (del 5q) cytogenetic abnormality received a single 10 mg oral dose of lenalidomide on Day -7 in the Pharmacokinetic Phase.
  During the Monotherapy Phase participants received 10 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg of lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
Period: Pharmacokinetic Phase
Arm/Group | 10 mg Non-del 5q | 15 mg Non-del 5q | 10 mg Del 5q
Started | 9 | 0 | 3
Completed | 8 | 0 | 3
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Monotherapy Phase
Arm/Group | 10 mg Non-del 5q | 15 mg Non-del 5q | 10 mg Del 5q
Started | 17 (Includes 8 participants from the PK Phase and 9 newly enrolled participants.) | 15 (All 15 participants were newly enrolled into the Monotherapy Phase.) | 7 (Includes 3 participants from the PK Phase and 4 newly enrolled participants.)
Safety Population | 17 (All patients who took at least 1 dose of study drug during Monotherapy or Combined Treatment Phase.) | 15 (All patients who took at least 1 dose of study drug during Monotherapy or Combined Treatment Phase.) | 7 (All patients who took at least 1 dose of study drug during Monotherapy or Combined Treatment Phase.)
Pharmacokinetic Population | 17 | 0 (Patients in the 15 mg Non-del 5q group were not included in the pharmacokinetic assessment.) | 7
Completed | 0 | 0 | 0
Not Completed | 17 | 15 | 7
Not completed — Adverse Event | 3 | 2 | 0
Not completed — Lack of therapeutic effect | 9 | 6 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other | 3 | 4 | 2
Period: Combined Treatment Phase
Arm/Group | 10 mg Non-del 5q | 15 mg Non-del 5q | 10 mg Del 5q
Started | 9 (Patients who discontinued the Monotherapy Phase due to erythroid non-response or erythroid relapse.) | 10 (Patients who discontinued the Monotherapy Phase due to erythroid non-response or erythroid relapse.) | 4 (Patients who discontinued the Monotherapy Phase due to erythroid non-response or erythroid relapse.)
Completed | 0 | 0 | 0
Not Completed | 9 | 10 | 4
Not completed — Lack of therapeutic effect | 8 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Non-del 5q | 15 mg Non-del 5q | 10 mg Del 5q | Total
Number analyzed (Participants) | 17 | 15 | 7 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.96) | 73.4 (6.51) | 72.6 (7.39) | 70.8 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 14 | 11 | 3 | 28
Race/Ethnicity, Customized [Number; unit: participants] — Participants could select more than 1 race option.
  participants
    White | 17 | 13 | 7 | 37
    Hispanic | 1 | 1 | 0 | 2
    Other | 1 | 1 | 0 | 2
Duration of MDS [Mean (Standard Deviation); unit: years] | 2.8 (2.28) | 2.6 (2.22) | 4.2 (4.74) | 3.0 (2.81)
International Prognostic Scoring System (IPSS) Score [Number; unit: participants] — The MDS IPSS score = sum of marrow blast + karyotype + cytopenia score. Score ranges from 0 (low risk) to 3.5 (high risk).
  participants
    Low risk (0) | 8 | 8 | 2 | 18
    Intermediate-1 (0.5-1.0) | 9 | 7 | 5 | 21
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status: 0 = Fully active, no restrictions; 1 = Restricted but ambulatory and capable of light work; 2 = Ambulatory and capable of self-care but unable to work.
  participants
    0 | 2 | 4 | 1 | 7
    1 | 14 | 11 | 6 | 31
    2 | 1 | 0 | 0 | 1
French-American-British (FAB) classification of MDS [Number; unit: participants] — Refractory anemia: characterized by less than 5% primitive blood cells (myeloblasts) in the bone marrow and pathological abnormalities primarily seen in red cell precursors; RARS: distinguished by the presence of 15% or greater red cell precursors in the marrow being abnormal iron-stuffed cells called "ringed sideroblasts"; RAEB: characterized by 5-20% myeloblasts in the marrow; RAEB-1: characterized by 5% to 9% blasts in the bone marrow and less than 5% blasts in the blood.
  participants
    Refractory anemia (RA) | 6 | 7 | 2 | 15
    Refractory anemia with ringed sideroblasts (RARS) | 5 | 6 | 0 | 11
    Refractory anemia with excess blasts (RAEB) | 3 | 1 | 4 | 8
    Refractory anemia with excess blasts -1 (RAEB-1) | 0 | 1 | 0 | 1
    Other | 3 | 0 | 1 | 4
Serum erythropoietin level [Number; unit: participants]
  < 500 mIU/mL | 9 | 4 | 2 | 15
  ≥ 500 mIU/mL | 7 | 2 | 5 | 14
  Missing | 1 | 9 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: PK Phase: Area-under-the Concentration-time Curve (AUC0-24) for Lenalidomide
Description: Area under the plasma concentration-time curve from Time 0 to 24 hours post-dose for lenalidomide after a single dose, calculated using the log-linear trapezoidal method.
Time Frame: On Day -7 blood samples were taken at predose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours post-dose.
Population: All Pharmacokinetic Phase participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 10 mg Lenalidomide: Participants received a single oral dose of 10 mg lenalidomide on Day -7.
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 12
ng*h/mL | 817 (30.5)

2. Secondary Outcome: PK Phase: Maximum Plasma Concentration of Lenalidomide (Cmax)
Description: The maximum observed plasma concentration (Cmax) of lenalidomide (its R- and S- enantiomers and the enantiomers combined) after a single dose on day -7.
Time Frame: On Day -7 blood samples were taken at predose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose.
Population: All Pharmacokinetic Phase participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 12
ng/mL
  Total Lenalidomide | 179 (33.6)
  S-Lenalidomide | 101 (34.9)
  R-Lenalidomide | 78.3 (32.7)

3. Secondary Outcome: Monotherapy Phase: Maximum Plasma Concentration of Lenalidomide (Cmax)
Description: The Maximum observed plasma concentration (Cmax) of lenalidomide (its R- and S- enantiomers and the enantiomers combined) after multiple dosing for 14 days.
Time Frame: On Day 14 blood samples were taken at predose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, and 5 hours postdose.
Population: Monotherapy Phase pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 10 mg Lenalidomide: During the Monotherapy Phase participants received 10 mg oral lenalidomide once daily.
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 24
ng/mL
  Total Lenalidomide | 185 (38.7)
  S-Lenalidomide | 104 (39)
  R-Lenalidomide | 80.7 (38.8)

4. Secondary Outcome: PK Phase: Terminal Half-life (t1/2)
Description: The apparent terminal half-life is the time required for plasma concentration to decrease by 50% after pseudo-equilibrium of distribution has been reached, and calculated as the natural logarithm of 2 (0.693) / Apparent terminal rate constant (λz).
Time Frame: as for outcome 2
Population: Pharmacokinetic Phase participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 12
hours
  Total Lenalidomide | 3.72 (19.5)
  S-Lenalidomide | 4.14 (29.0)
  R-Lenalidomide | 3.58 (21.4)

5. Secondary Outcome: PK Phase: Percent of Administered Lenalidomide Excreted Over 24 Hours After a Single, Oral Dose
Description: Percent of the administered dose of lenalidomide excreted unchanged in urine over 24 hours postdose after a single dose on Day -7, calculated as:
  (amount excreted unchanged in urine over 24 hours postdose / Dose) * 100.
  The dose was 10 mg for total lenalidomide and 5 mg for the enantiomers.
Time Frame: On Day -7 at predose and over the intervals of 0-5, 5-8, 8-12, and 12-24 hours postdose.
Population: PK Phase participants for whom data was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent of administered dose
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 8
percent of administered dose
  Total Lenalidomide | 65.1 (13.5)
  S-Lenalidomide | 67.9 (13.9)
  R-Lenalidomide | 62.2 (14.0)

6. Secondary Outcome: Monotherapy Phase: Percent of Lenalidomide Excreted Over 5 Hours Post Day 14 Dose
Description: Percent of the administered lenalidomide dose excreted unchanged in urine over 5 hours postdose after multiple dosing for 14 days, calculated as:
  (amount excreted unchanged in urine over the first 5 hours postdose / Dose) * 100.
  The dose was 10 mg for total lenalidomide and 5 mg for the enantiomers.
Time Frame: On Day 14, at predose and over the interval of 0-5 hours postdose.
Population: Monotherapy Phase Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent of administered dose
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 24
percent of administered dose
  Total Lenalidomide | 34.0 (60.3)
  S-Lenalidomide | 35.4 (59.0)
  R-Lenalidomide | 32.5 (62.0)

7. Secondary Outcome: Time to Grade 4 Neutropenia or Thrombocytopenia
Description: Time to the first event of grade 4 neutropenia or thrombocytopenia, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0, was calculated as date of first event - date of first dose + 1.
Time Frame: From the date of first dose until 30 days after the last dose (up to 1218 days)
Population: Safety population, which comprised all enrolled patients who took at least 1 dose of study drug during the Monotherapy Phase or the Combined Treatment Phase.
Measure: Median (Full Range); unit: days
Groups:
- Non-del 5q: Participants with low- or intermediate-1-risk myelodysplastic syndromes (MDS) not associated with a deletion 5q (del 5q) cytogenetic abnormality received 10 or 15 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  During the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
- Del 5q: Participants with a deletion 5q (del 5q) cytogenetic abnormality received 10 mg oral lenalidomide once daily in the Monotherapy Phase. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  During the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg of lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
Arm/Group | Non-del 5q | Del 5q
Number analyzed (Participants) | 32 | 7
days
  Grade 4 Neutropenia | 69.0 [11 to 168] | 28.0 [17 to 36]
  Grade 4 Thrombocytopenia | 53.0 [22 to 141] | 29.0 [22 to 36]

8. Secondary Outcome: Percentage of Participants With a Erythroid Response Across All Phases
Description: Erythroid response was categorized as either a major response or a minor response. A major response was defined as red blood cell (RBC) transfusion independence during any consecutive 56-day period and an increase in hemoglobin of at least 1.5 g/dL. A minor response was defined as a ≥ 50% or ≥ 4 unit decrease in RBC transfusions from pretreatment requirements (the number of RBC transfusions required over an 8-week period before the start of study drug treatment).
Time Frame: Assessed every 28 days until study discontinuation (up to 1218 days).
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Non-del 5q | 15 mg Non-del 5q | 10 mg Del 5q
Number analyzed (Participants) | 17 | 15 | 7
percentage of participants
  Major response | 17.6 | 40.0 | 85.7
  Minor response | 5.9 | 0 | 0

9. Secondary Outcome: Percentage of Participants Overall With Erythroid Response by Baseline Erythropoietin Level
Description: To evaluate the predictive value of pretreatment serum erythropoietin (EPO) concentration for erythroid response to lenalidomide, the percentage of erythroid responders versus non-responders were stratified by Baseline EPO levels (≤ 500 mIU/mL versus > 500 mIU/mL). Response includes participants with either a major or minor response.
Time Frame: Assessed every 28 days until study discontinuation (up to 1218 days)
Population: Safety population.
Measure: Number; unit: percentage of participants
Groups:
- Responders: Participants with a erythroid response.
- Non-responders: Participants who were not erythroid responders.
- Overall: All participants in the Safety population.
Arm/Group | Responders | Non-responders | Overall
Number analyzed (Participants) | 16 | 23 | 39
percentage of participants
  Baseline EPO ≤ 500 mIU/mL | 62.5 | 47.8 | 53.8
  Baseline EPO > 500 mIU/mL | 37.5 | 39.1 | 38.5

10. Secondary Outcome: Change From Baseline in Bone Marrow Cellularity and Correlation With Grade 4 Myelosuppression
Description: Bone marrow cellularity is the volume ratio of hematopoietic stem cells and adipocytes (fat cells). Due to the small number of bone marrow samples, this analysis was not performed.
Time Frame: Baseline and Week 16
Population: Unable to obtain sufficient bone marrow samples to perform analyses.
Groups:
- Non-del 5q: Participants with low- or intermediate-1-risk myelodysplastic syndromes (MDS) not associated with a deletion 5q (del 5q) cytogenetic abnormality received 10 or 15 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
- Del 5q: Participants with a deletion 5q (del 5q) cytogenetic abnormality received 10 mg oral lenalidomide once daily in the Monotherapy Phase. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg of lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
Arm/Group | Non-del 5q | Del 5q
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Monotherapy Phase: Area-under-the Concentration-time Curve (AUC0-5) for Lenalidomide
Description: Area under the plasma concentration-time curve from Time 0 to 5 hours postdose for lenalidomide (its R- and S- enantiomers and the enantiomers combined) after multiple dosing for 14 days, calculated using the log-linear trapezoidal method.
Time Frame: On Day 14 blood samples were taken at predose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, and 5 hours postdose.
Population: Monotherapy Phase pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Lenalidomide
Number analyzed (Participants) | 24
ng*h/mL
  Total Lenalidomide | 563 (32.5)
  S-Lenalidomide | 315 (34.2)
  R-Lenalidomide | 248 (30.6)

12. Secondary Outcome: Marrow-infiltrating Lymphocyte (MIL) Number and Cytolytic Activity
Description: Due to the low number of bone marrow samples collected this analysis was not performed.
Time Frame: Pre-Study and Week 16
Population: Unable to obtain sufficient bone marrow samples to perform analyses
Arm/Group | Non-del 5q | Del 5q
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The safety analyses were conducted on data collected from the time of first dose of study drug to 30 days after the last dose of study drug.
Groups:
- 10 mg Lenalidomide: Participants with low- or intermediate-1-risk myelodysplastic syndromes (MDS) received a single 10 mg oral dose of lenalidomide on Day -7 in the Pharmacokinetic Phase.
  During the Monotherapy Phase participants received 10 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 10 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
- 15 mg Lenalidomide: Participants with low- or intermediate-1-risk MDS were enrolled directly into the Monotherapy Phase and received 15 mg oral lenalidomide once daily. Erythroid responders could continue lenalidomide monotherapy in the absence of limiting toxicity, disease progression, or erythroid failure.
  After the completion of 16 weeks of lenalidomide monotherapy, in the Combined Treatment Phase participants who were erythroid nonresponders and erythroid responders who had developed an erythroid relapse continued treatment with 15 mg lenalidomide daily in conjunction with recombinant human erythropoietin (rhu EPO) 40,000 units administered weekly by subcutaneous injection for 8 weeks. Responding patients could continue combined treatment.
Arm/Group | 10 mg Lenalidomide | 15 mg Lenalidomide
Serious Adverse Events (participants affected / at risk) | 10/24 | 5/15
Other Adverse Events (participants affected / at risk) | 24/24 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Lenalidomide (N=24) | 15 mg Lenalidomide (N=15)
Asthenia (General disorders) | 0 | 1
Disease progression NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 1
Parotitis (Infections and infestations) | 1 | 0
Sepsis NOS (Infections and infestations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Gangrene NOS (Vascular disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Lenalidomide (N=24) | 15 mg Lenalidomide (N=15)
Neutropenia (Blood and lymphatic system disorders) | 22 | 14
Leukopenia NOS (Blood and lymphatic system disorders) | 21 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 11
Anaemia NOS (Blood and lymphatic system disorders) | 17 | 9
Autoimmune haemolytic anaemia NOS (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea NOS (Gastrointestinal disorders) | 10 | 11
Constipation (Gastrointestinal disorders) | 5 | 5
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 1 | 4
Vomiting NOS (Gastrointestinal disorders) | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Loose stools (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 7
Rash NOS (Skin and subcutaneous tissue disorders) | 7 | 2
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 | 3
Contusion (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis NOS (Skin and subcutaneous tissue disorders) | 1 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 6 | 4
Pyrexia (General disorders) | 6 | 2
Asthenia (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 3 | 2
Pain NOS (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Gait abnormal (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection NOS (Infections and infestations) | 5 | 3
Urinary tract infection NOS (Infections and infestations) | 0 | 4
Sinusitis NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Tooth infection (Infections and infestations) | 1 | 2
Ear infection NOS (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 1
Body tinea (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 0 | 1
Otitis externa NOS (Infections and infestations) | 0 | 1
Respiratory tract infection NOS (Infections and infestations) | 0 | 1
Vaginitis bacterial NOS (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 1 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Sleep apnoea syndrome (Nervous system disorders) | 0 | 1
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 4
Appetite decreased NOS (Metabolism and nutrition disorders) | 1 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Blood in stool (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Computerised tomogram abnormal (Investigations) | 0 | 1
Faecal occult blood positive (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Vitamin b12 decreased (Investigations) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Pallor (Vascular disorders) | 0 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Deafness NOS (Ear and labyrinth disorders) | 0 | 1
Acquired hypothyroidism (Endocrine disorders) | 0 | 1
Hypersensitivity NOS (Immune system disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication. It has priority over subset (single center) publication, for duration of 1 year after study completion.
* Individual investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 60 days.